CLINICAL TRIAL: NCT06025903
Title: Assessing the Role of Mitochondrial Dysfunction in Primary Progressive Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Azienda Socio Sanitaria Territoriale della Valle Olona (Other)
Responsible Party: Principal Investigator, Melissa Sorosina, Principal Investigator, IRCCS San Raffaele
Other Study IDs: MitoMS_GR-2019-12368672
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; mitochondria
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Progressive multiple sclerosis: patients affected by primary progressive multiple sclerosis
- Relapsing Remitting multiple sclerosis: patients affected by primary progressive multiple sclerosis

SUMMARY:
The purpose of this project is to study genetic determinants of mitochondrial impairment in primary progressive multiple sclerosis. Specific aims are: 1) identify mitochondrial-related pathways, inherited and somatic mitochondrial DNA mutations associated to primary progressive multiple sclerosis, 2) functionally assess the identified genetic alterations.

DETAILED DESCRIPTION:
Multiple Sclerosis is a major cause of neurological disability, with a high socio-economic impact that increases as disability progresses. Effective treatment of primary progressive multiple sclerosis is still an unmet need and the underlying neurodegenerative processes have to be fully investigated. The purpose of this project is to study genetic determinants of mitochondrial impairment in primary progressive multiple sclerosis. Altered mitochondrial pathways will be investigate, as well as inherited and tissue-specific somatic mitochondrial variations associated with primary progressive multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by primary progressive or relapsing remitting multiple sclerosis
* Patient able to provide informed consent

Exclusion Criteria:

* Individuals with < 18 years
* Patients not affected by primary progressive or relapsing remitting multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be recruited from primary care clinic
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
sequencing of mitochondrial DNA | 3 years
  the mitochondrial DNA collected from blood and cerebrospinal fluid will be sequenced and analysed, comparing the frequency of variants between the two disease courses

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Sorosina, Principal Investigator — IRCCS San Raffaele
Locations (2):
- Italy (2):
  - IRCCS San Raffaele, Milan, MI
  - ASST della Valle Olona - Ospedale di Gallarate, Gallarate, VA

IPD SHARING:
Plan to Share IPD: No